CLINICAL TRIAL: NCT02152163
Title: Assessing the Efficacy of IV Ibuprofen for Treatment of Pain in Orthopedic Trauma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Delray Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: WIRB Protocol #20121749
Record Dates: First submitted 2014-05-16; First posted 2014-06-02 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Pain
Keywords: Ibuprofen; Caldolor; orthopedic trauma
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: , randomized, double-blind, parallel-group, placebo-controlled study. Eligible patients who signed the informed consent were randomized to either IV Ibuprofen (Caldolor®) or Placebo via a computer-generated randomization list.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Staff, including the principal investigator, study coordinator, and trauma nurses and the patients were blinded as to the treatment they received. In order to maintain the double-blind protocol, all IV bags had identical appearance and label.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Ibuprofen 800 mg (Active Comparator): IV Ibuprofen 800 mg
  Interventions: Drug: IV Ibuprofen
- IV Saline (Placebo Comparator): IV Saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IV Ibuprofen
  Other Names: IV Caldolor
  Arms: IV Ibuprofen 800 mg
Drug: placebo
  Other Names: iv saline
  Arms: IV Saline

SUMMARY:
STUDY OBJECTIVES:

1. To evaluate the effectiveness of around the clock (OTC) IV ibuprofen (8 doses) in decreasing pain in orthopedic trauma patients with fractures of the extremities, face, pelvis and/or ribs compared to patients not receiving the medication.
2. To evaluate the effectiveness of around the clock (OTC) IV ibuprofen (8 doses) in decreasing the use of opioid analgesics among orthopedic trauma patients with fractures of the extremities, face, pelvis, and/or ribs compared to compared to patients not receiving the medication.

DETAILED DESCRIPTION:
Eligible patients were trauma patients between the ages of 18 and 75 years old with adequate IV access who were able to self-report and communicate pain severity and who were consecutively admitted to the trauma intensive care unit (ICU) or trauma step-down units with a fracture of the ribs, face, extremities and/or pelvis.

Eligible patients who signed the informed consent were randomized to either IV Ibuprofen (Caldolor®) or Placebo via a computer-generated randomization list.

Patients had pain measured using a Numerical Rating Scale (NRS) that ranged from 0 (no pain) to 10 (worst possible pain)

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patient admitted to Trauma ICU or Trauma Step-Down Units.
2. Fracture of ribs, face, extremities and/or pelvis
3. Age between 18 and 75 years old
4. Adequate IV access
5. Able to self report and communicate pain severity

Exclusion Criteria:

1. History of allergy or hypersensitivity to any component of IV Ibuprofen, aspirin (or aspirin related products) NSAIDs, or COX-2 inhibitors
2. Any intracranial or spinal cord trauma
3. History of clinically significant bleeding disorders including ITP, DIC or platelet dysfunction
4. Recent history of intracranial surgery or stroke (within past 30 days)
5. History of ulcers, gastritis or previous GI bleeding
6. Renal Impairment (Creatinine > 3.0 mg/dL)
7. Pregnant or breastfeeding
8. Otherwise unsuitable in the opinion of the treating physician at time of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Weisz, MD, Principal Investigator — Delray Medical Center
Locations (1):
- Delray Medical Center, Delray Beach, Florida, United States

REFERENCES:
- [Background] Bayouth L, Safcsak K, Cheatham ML, Smith CP, Birrer KL, Promes JT. Early intravenous ibuprofen decreases narcotic requirement and length of stay after traumatic rib fracture. Am Surg. 2013 Nov;79(11):1207-12. PMID 24165259
- [Background] Drendel AL, Lyon R, Bergholte J, Kim MK. Outpatient pediatric pain management practices for fractures. Pediatr Emerg Care. 2006 Feb;22(2):94-9. doi: 10.1097/01.pec.0000199564.64264.f4. PMID 16481924
- [Result] Weisz RD, Fokin AA, Lerner V, Flynt A, Macias-Perez I, Pavliv L, Crawford M, Puente I. Intravenous Ibuprofen Reduces Opioid Consumption During the Initial 48 Hours After Injury in Orthopedic Trauma Patients. J Orthop Trauma. 2020 Jul;34(7):341-347. doi: 10.1097/BOT.0000000000001733. PMID 31929374

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Ibuprofen 800 mg: IV Ibuprofen 800 mg
  IV Ibuprofen
- IV Saline: IV Saline
  placebo
Period: Overall Study
Arm/Group | IV Ibuprofen 800 mg | IV Saline
Started | 51 | 48
Completed | 39 | 35
Not Completed | 12 | 13
Not completed — Physician Decision | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ibuprofen 800 mg | IV Saline | Total
Number analyzed (Participants) | 39 | 35 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 35 | 74
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 30 | 28 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 35 | 74

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of IV Ibuprofen in Orthropedic Trauma Patients
Description: Outcome measure based on morphine equivalent dosage comparing the two groups
Time Frame: morphine equivalent dosage in over 48 hours after admission
Measure: Least Squares Mean (95% Confidence Interval); unit: morphine equivalent dosage, mg
Arm/Group | IV Ibuprofen 800 mg | IV Saline
Number analyzed (Participants) | 39 | 35
morphine equivalent dosage, mg | 74.9 [62.1 to 87.8] | 97.8 [84.4 to 111.2]

ADVERSE EVENTS:
Time Frame: 3 years
Description: No adverse events identified
Arm/Group | IV Ibuprofen 800 mg | IV Saline
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/35
Other Adverse Events (participants affected / at risk) | 0/39 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-06-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT02152163/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT02152163/SAP_001.pdf